CLINICAL TRIAL: NCT02290873
Title: A Prospective, Double-blind, Randomized, Placebo and Active Controlled, Multi-center, Parallel Group Study Comparing Remimazolam to Placebo, With an Additional Open-label Arm For Midazolam, in Patients Undergoing a Colonoscopy
Brief Title: A Phase III Study of the Efficacy and Safety of Remimazolam Compared to Placebo and Midazolam in Colonoscopy Patients
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Paion UK Ltd. (Industry)
Collaborators: Premier Research (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CNS7056-006
Record Dates: First submitted 2014-11-07; First posted 2014-11-14 (Estimated); Results first posted 2018-11-09 (Actual); Last update posted 2020-10-20 (Actual); Status verified 2020-09

CONDITIONS: Colonoscopy
MeSH Terms: interventions — remimazolam; Midazolam

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Remimazolam (Experimental): Remimazolam iv 5 mg for sedation induction, and 2.5 mg top-ups for sedation maintenance.
  Fentanyl pre-treatment: 50 μg (or less for elderly/disabled subjects) and 25 μg top-up doses
  Interventions: Drug: Remimazolam
- Placebo (Placebo Comparator): Inactive control arm
  Fentanyl pre-treatment: 50 μg (or less for elderly/disabled subjects) and 25 μg top-up doses
  Interventions: Drug: Placebo
- Midazolam (Active Comparator): Midazolam iv 1.75 mg* for sedation induction and 1.0 mg* for sedation maintenance.
  *1.0 mg for induction and 0.5 mg for maintenance in adults over 60, debilitated or chronically ill
  Fentanyl pre-treatment: 50 μg (or less for elderly/disabled subjects) and 25 μg top-up doses
  Interventions: Drug: Midazolam

INTERVENTIONS:
Drug: Remimazolam — For induction and maintenance of sedation
  Other Names: Byfavo, CNS7056
  Arms: Remimazolam
Drug: Midazolam — For induction of maintenance and sedation
  Other Names: Versed
  Arms: Midazolam
Drug: Placebo — Inactive control arm
  Arms: Placebo

SUMMARY:
A prospective, double-blind, randomized, placebo and active controlled, multi-center, parallel group study comparing remimazolam to placebo, with an additional open-label arm for midazolam, in patients undergoing a colonoscopy for diagnostic or therapeutic reasons.

ELIGIBILITY:
Inclusion Criteria:

* Male and female patients, aged ≥18, scheduled to undergo a diagnostic or therapeutic colonoscopy (therapeutic procedures could include hemostasis, resection, ablation decompression, foreign body extraction, for example).
* American Society of Anesthesiologists Score 1 through 3
* Body mass index ≤40 kg/m2.
* For female patients with child-bearing potential, negative result of pregnancy test (serum or urine) as well as use of birth control during the study period (from the time of consent until all specified observations were completed).
* Patient voluntarily signed and dated an informed consent form that was approved by an Independent Review Board prior to the conduct of any study procedure.
* Patient was willing and able to comply with study requirements and return for a Follow-up Visit on Day 4 (+3/-1 days) after the colonoscopy.

Exclusion Criteria:

* Patients with a known sensitivity to benzodiazepines, flumazenil, opioids, naloxone, or a medical condition such that these agents were contraindicated.
* Chronic use of benzodiazepines for any indication (eg, insomnia, anxiety, spasticity).
* Chronic use of opioids for any indication.
* Female patients with a positive serum human chorionic gonadotropin pregnancy test at screening or baseline.
* Lactating female patients.
* Patients with positive drugs of abuse screen or a positive serum ethanol at baseline.
* Patient with a history of drug or ethanol abuse within the past 2 years.
* Patients in receipt of any investigational drug within 30 days or less than seven half-lives (whichever was longer) before screening, or scheduled to receive one during the study period.
* Participation in any previous clinical trial with remimazolam.
* Patients with an inability to communicate well in English with the investigator, or deemed unsuitable according to the investigator (in each case providing a reason).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 461 (Actual)
Dates: Start 2015-03-30 (Actual); Primary Completion 2016-04 (Actual); Study Completion 2016-04-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Douglas K Rex, MD, Principal Investigator — Indiana University School of Medicine
Locations (13):
- United States (13):
  - University of South Alabama, Mobile, Alabama
  - Advanced Clinical Research Institute, Anaheim, California
  - Precision Research Institute, Chula Vista, California
  - Precision Research Institute, San Diego, California
  - Borland-Grover Clinic, P.A, Jacksonville, Florida
  - Indiana University Health, Indianapolis, Indiana
  - Delta Research Partners Inc, Monroe, Louisiana
  - Washington University School of Medicine, St Louis, Missouri
  - Wake Research Associates, Raleigh, North Carolina
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - Thomas Jefferson Medical College, Philadelphia, Pennsylvania
  - Nashville Medical Research Institute, Nashville, Tennessee
  - Gastroenterology Associates of Tidewater, Chesapeake, Virginia

REFERENCES:
- [Background] Antonik LJ, Goldwater DR, Kilpatrick GJ, Tilbrook GS, Borkett KM. A placebo- and midazolam-controlled phase I single ascending-dose study evaluating the safety, pharmacokinetics, and pharmacodynamics of remimazolam (CNS 7056): Part I. Safety, efficacy, and basic pharmacokinetics. Anesth Analg. 2012 Aug;115(2):274-83. doi: 10.1213/ANE.0b013e31823f0c28. Epub 2011 Dec 20. PMID 22190555
- [Background] Wiltshire HR, Kilpatrick GJ, Tilbrook GS, Borkett KM. A placebo- and midazolam-controlled phase I single ascending-dose study evaluating the safety, pharmacokinetics, and pharmacodynamics of remimazolam (CNS 7056): Part II. Population pharmacokinetic and pharmacodynamic modeling and simulation. Anesth Analg. 2012 Aug;115(2):284-96. doi: 10.1213/ANE.0b013e318241f68a. Epub 2012 Jan 16. PMID 22253270
- [Background] Worthington MT, Antonik LJ, Goldwater DR, Lees JP, Wilhelm-Ogunbiyi K, Borkett KM, Mitchell MC. A phase Ib, dose-finding study of multiple doses of remimazolam (CNS 7056) in volunteers undergoing colonoscopy. Anesth Analg. 2013 Nov;117(5):1093-100. doi: 10.1213/ANE.0b013e3182a705ae. PMID 24108261
- [Background] Borkett KM, Riff DS, Schwartz HI, Winkle PJ, Pambianco DJ, Lees JP, Wilhelm-Ogunbiyi K. A Phase IIa, randomized, double-blind study of remimazolam (CNS 7056) versus midazolam for sedation in upper gastrointestinal endoscopy. Anesth Analg. 2015 Apr;120(4):771-80. doi: 10.1213/ANE.0000000000000548. PMID 25502841
- [Background] Pambianco DJ, Borkett KM, Riff DS, Winkle PJ, Schwartz HI, Melson TI, Wilhelm-Ogunbiyi K. A phase IIb study comparing the safety and efficacy of remimazolam and midazolam in patients undergoing colonoscopy. Gastrointest Endosc. 2016 May;83(5):984-92. doi: 10.1016/j.gie.2015.08.062. Epub 2015 Sep 9. PMID 26363333
- [Result] Douglas K. Rex, MD, MACG, Raj Bhandari, MD, Taddese Desta MD, Michael DeMicco MD, Cynthia Schaeffer MD, Kyle Etzkorn, Charles Barish MD, Ronald Pruitt MD, Brooks Cash MD, FACG, Daniel Quirk MD, Felix Tiongco MD, David Bernstein MD, FACG. REMIMAZOLAM IS A SAFE AND EFFECTIVE AGENT FOR SEDATION IN OUTPATIENT COLONOSCOPY: RESULTS OF A PHASE 3, MULTICENTER, RANDOMIZED, PLACEBO CONTROLLED TRIAL. Program No. ACG 2016 Annual Scientific Meeting Abstracts. Las Vegas, NV: American College of Gastroenterology.
- [Result] Rex DK, Bhandari R, Desta T, DeMicco MP, Schaeffer C, Etzkorn K, Barish CF, Pruitt R, Cash BD, Quirk D, Tiongco F, Sullivan S, Bernstein D. A phase III study evaluating the efficacy and safety of remimazolam (CNS 7056) compared with placebo and midazolam in patients undergoing colonoscopy. Gastrointest Endosc. 2018 Sep;88(3):427-437.e6. doi: 10.1016/j.gie.2018.04.2351. Epub 2018 Apr 30. PMID 29723512

RESULTS

PARTICIPANT FLOW:
Groups:
- Remimazolam: Double-blind Remimazolam iv arm: 5 mg for sedation induction, and 2.5 mg top-ups for sedation maintenance.
- Placebo: Double-blind Placebo iv arm: as an inactive control
- Midazolam: Open-label Midazolam iv arm: 1.75 mg* for sedation induction and 1.0 mg* for sedation maintenance.
  *1.0 mg for induction and 0.5 mg for maintenance in adults over 60, debilitated or chronically ill
Period: Overall Study
Arm/Group | Remimazolam | Placebo | Midazolam
Started | 298 | 60 | 103
Modified Intention to Treat (mITT) (All ITT population who received at least 1 complete dose of study medication) | 296 | 60 | 102
Safety Population (All randomized patients who received any amount of study drug and were analyzed as treated) | 296 | 60 | 102
Completed | 296 | 59 | 101
Not Completed | 2 | 1 | 2
Not completed — Withdrawal by Subject | 0 | 1 | 1
Not completed — Nellcor device error | 1 | 0 | 0
Not completed — Esophagogastroduodenoscopy was added | 1 | 0 | 0
Not completed — Protocol Violation | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: Baseline Analysis Population is the safety population
Groups:
- Placebo: Double-blind Placebo iv arm: inactive control arm
- Total: Total of all reporting groups
Arm/Group | Remimazolam | Placebo | Midazolam | Total
Number analyzed (Participants) | 296 | 60 | 102 | 458
Age, Continuous [Mean (Standard Deviation); unit: years] | 54.4 (10.12) | 56 (9.51) | 55.6 (10.15) | 54.9 (10.05)
Age, Customized [Count of Participants; unit: Participants]
  <65 years | 254 | 53 | 88 | 395
  ≥65 years | 42 | 7 | 14 | 63
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 149 | 35 | 56 | 240
  Male | 147 | 25 | 46 | 218
Region of Enrollment [Number; unit: participants]
  United States | 296 | 60 | 102 | 458
Weight [Mean (Standard Deviation); unit: Kg] | 83.2 (17.39) | 84.6 (19.9) | 81.9 (16.24) | 83.1 (17.47)
Height [Mean (Standard Deviation); unit: cm] | 170.1 (10.36) | 167.8 (10.24) | 169.5 (11.15) | 169.6 (10.53)
Body Max Index (BMI) [Mean (Standard Deviation); unit: kg/m2] | 28.9 (4.72) | 30 (5.31) | 28.8 (4.75) | 29 (4.81)

OUTCOME MEASURES:

1. Primary Outcome: Success Rates of the Procedure
Description: Success of the Procedure is measured by completion of colonoscopy, no requirement for an alternative sedative and no requirement for more than 5 top-ups of study medication within any 15 minute period in the blinded arms (remimazolam/placebo) or no requirement for more than 3 doses within any 12 minute window in the midazolam arm.
Time Frame: From administration of the first dose of the study drug to the end of colonoscopy
Measure: Count of Participants; unit: Participants
Groups:
- Placebo: Double-blind Placebo iv arm: as an inactive control arm
Arm/Group | Remimazolam | Placebo | Midazolam
Number analyzed (Participants) | 298 | 60 | 103
Participants | 272 | 1 | 26
Statistical Analysis 1: Comparison: Remimazolam vs Placebo; Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel — P-value calculated from a Cochran-Mantel-Haenszel test accounting for fentanyl strata; Difference in Rates = 0.8961, 95% CI 2-sided [0.8505 to 0.9416]

2. Secondary Outcome: Time to Start of Procedure
Description: The time to the start of the procedure after administration of the first dose of randomized study drug
Time Frame: From first dose of study drug until insertion of the colonoscope
Population: Patients who do not reach the endpoint are excluded from the analysis.
Measure: Median (Inter-Quartile Range); unit: minutes
Arm/Group | Remimazolam | Placebo | Midazolam
Number analyzed (Participants) | 296 | 60 | 102
minutes | 4 [3.0 to 6.0] | 19.5 [17.0 to 23.0] | 19 [12.0 to 21.0]
Statistical Analysis 1: Comparison: Remimazolam vs Placebo; Test type: Superiority; p < 0.0001, Log Rank; Hazard Ratio (HR) = 6.133, 95% CI 2-sided [4.416 to 8.517]

3. Secondary Outcome: Time to Fully Alert
Description: The time to fully alert (time to first of three consecutive Modified Observer's Assessment of Alertness/Sedation [MOAA/S] scores of 5) after the end of colonoscopy procedure [colonoscope out], and after the last dose of study drug or rescue sedative medication
Time Frame: From the end of colonoscopy (colonoscope out) until the patient has recovered to fully alert and from the last injection of the study drug or rescue sedative medication until the patient has recovered to fully alert
Population: Patients who do not reach the endpoint are censored at last MOAA/S
Measure: Median (95% Confidence Interval); unit: minutes
Arm/Group | Remimazolam | Placebo | Midazolam
Number analyzed (Participants) | 296 | 60 | 102
minutes
  After the end of colonoscopy: number analyzed (Participants) | 293 | 59 | 101
  After the end of colonoscopy | 6 [5 to 7] | 15 [13 to 21] | 13 [11 to 16]
  After last dose of study drug or rescue sedative | 14 [13 to 14] | 28 [24 to 32] | 24 [22 to 26]

4. Secondary Outcome: Time to Ready for Discharge
Description: The time after the end of colonoscopy procedure (colonoscope out) and after the last injection of study drug or rescue sedative medication, until discharge (defined as ability to walk unassisted).
Time Frame: From the end of the colonoscopy until discharge (expected to be the same day). After the last dose of study drug or rescue sedative, until discharge (expected to be the same day).
Measure: Median (95% Confidence Interval); unit: minutes
Arm/Group | Remimazolam | Placebo | Midazolam
Number analyzed (Participants) | 296 | 60 | 102
minutes
  After the end of colonoscopy procedure | 44 [42 to 46] | 49 [44 to 54] | 48 [41 to 51]
  After last dose of study drug or rescue sedative | 51 [49 to 54] | 60.5 [55 to 67] | 57 [53 to 61]

ADVERSE EVENTS:
Time Frame: From first dose of study drug until Day 4, or resolution of any ongoing adverse events
Description: Total number of participants affected with Other (Not Including Serious) Adverse Events represents any participant in the trial with a non serious Treatment-emergent Adverse Event (TEAE). The listing of participants with Preferred Term (PT)TEAEs is reported with a threshold of 5% in any of the arms
Arm/Group | Remimazolam | Placebo | Midazolam
All-Cause Mortality (participants affected / at risk) | 0/296 | 0/60 | 0/102
Serious Adverse Events (participants affected / at risk) | 0/296 | 0/60 | 0/102
Other Adverse Events (participants affected / at risk) | 218/296 | 47/60 | 93/102
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Remimazolam (N=296) | Placebo (N=60) | Midazolam (N=102)
Hypotension (Vascular disorders) | 115 | 25 | 63
Hypertension (Vascular disorders) | 59 | 17 | 18
Bradycardia (Cardiac disorders) | 33 | 7 | 16
Diastolic Hypertension (Vascular disorders) | 29 | 6 | 9
Diastolic Hypotension (Vascular disorders) | 23 | 4 | 9
Systolic hypertension (Vascular disorders) | 16 | 5 | 6
Tachycardia (Cardiac disorders) | 23 | 7 | 13
Nausea (Gastrointestinal disorders) | 5 | 4 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
At least 60 days prior to submission of communications, sponsor shall review and comment on the communications. Sponsor shall have the right to require institution and investigator to remove specifically identified confidential information and to delay the proposed publication an additional 60 days to enable sponsor to seek patent protection.